CLINICAL TRIAL: NCT00518141
Title: Use of Acetylsalicylic Acid and Terbutalin in ART
Brief Title: Use of Acetyl Salicylic Acid and Terbutalin in Assisted Reproductive Techniques (ART)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset Telemark (Other Government)
Responsible Party: Jarl Kahn, Fertilitetsklinikken Sør
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-06085 (REK)
Record Dates: First submitted 2007-08-17; First posted 2007-08-20 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2011-07

CONDITIONS: Reproductive Techniques, Assisted
MeSH Terms: conditions — Helping Behavior | interventions — Terbutaline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Experimental): FER
  Interventions: Drug: Acetyl Salicylic Acid and Terbutalin
- 2 (No Intervention): FER
- 3 (Experimental): SET
  Interventions: Drug: Acetyl Salicylic Acid and Terbutalin
- 4 (No Intervention): SET
- 5 (Experimental): DET
  Interventions: Drug: Acetyl Salicylic Acid and Terbutalin
- 6 (No Intervention): DET

INTERVENTIONS:
Drug: Acetyl Salicylic Acid and Terbutalin — ASA 75 mg, Terbutalin 5mg
  Arms: 1; 3; 5

SUMMARY:
This study aims to determine the possible effects of Acetyl Salicylic Acid (ASA) and Terbutalin on ART treatment.

DETAILED DESCRIPTION:
This study aims to determine the possible effects of ASA and Terbutalin on ART treatment.

ELIGIBILITY:
Inclusion Criteria:

* Infertile women below 39 years of age

Exclusion Criteria:

* Women who may react allergically to the drugs administered
* Women with hyperthyroid or IDDM
* Women who do not want to participate in the study
* Women who are unable to give informed, written consent.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2006-03; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Pregnancy | 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jarl A Kahn, Dr. med, Principal Investigator — STHF, Kvinneklinikken, Fertilitetsklinikken Sor
Locations (1):
- STHF, Kvinneklinikken, Fertilitetsklinikken Sor, Porsgrunn, Telemark, Norway